CLINICAL TRIAL: NCT02615249
Title: Clinical Evaluation of Metal Panel Allergens: Aluminum, Copper, Manganese, Molybdenum, Tin, Titanium, Vanadium and Zinc Dose Response Study
Brief Title: Clinical Evaluation of Metal Panel Allergens: Dose Response Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allerderm (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SP148MP201
Record Dates: First submitted 2015-11-23; First posted 2015-11-26 (Estimated); Results first posted 2020-08-11 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-04

CONDITIONS: Dermatitis, Eczematous
MeSH Terms: conditions — Eczema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Metal Allergen Epicutaneous Patch (Experimental): 8 allergens were tested. Not all subjects tested each allergen. Section reports number of subjects with positive responses to each allergen.
  Interventions: Biological: Metal Allergen Epicutaneous Patch

INTERVENTIONS:
Biological: Metal Allergen Epicutaneous Patch — 48 hour application of metal allergen patch to diagnose contact dermatitis

SUMMARY:
48-hour application of metal allergen patches to test for potential allergic responses.

DETAILED DESCRIPTION:
A 48-hour application (approximate) of investigational allergen panels, excipient controls and corresponding reference allergens will be applied to the skin of human subjects to test for potential positive allergic responses. Test sites will be evaluated at 3-4, 7-8, 10-14 and 19-23 days after application. Ascending allergen dosages will be randomized within each panel into three different configurations which will be randomly assigned to subjects as they enter the study. The investigators and subjects will be aware of the allergens and the patch test doses but will not be aware of the location of individual allergens within each panel.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older.
2. Past positive patch test result within the past 10 years (to one of the dilution series metals being tested on this study) or strong suspicion of metal contact allergy based on results of the Qualification Questionnaire.
3. Unable to become pregnant or willing to use an acceptable method of contraception to prevent pregnancy if female of childbearing potential; (Inability to become pregnant includes all male subjects and female subjects who are postmenopausal for at least 1 year, or surgically sterile- have had a hysterectomy, bilateral ovariectomy, uterine ablation or bilateral tubal ligation. Acceptable methods of contraception include: 1) systemic birth control; 2) double barrier method; 3) intrauterine device; 4) vasectomized partner; or 5) abstinence from sexual intercourse. Subject must agree to use acceptable contraception for the duration of the entire study.)
4. Understands and signs the approved Informed Consent form which is consistent with all institutional, local and national regulations.

Exclusion Criteria:

1. Breastfeeding or pregnant (as determined by urine pregnancy test) or intending to become pregnant during the course of the study.
2. Topical treatment with corticosteroids or other immunosuppressive agents on or near the test area during the 14 days prior to inclusion in this study.
3. Systemic treatment with corticosteroids (equivalent to > 10 mg prednisone) or other immunosuppressive agents during the 14 days prior to inclusion in this study. Inhaled treatments are permitted. NOTE: Steroidal nose or eye drops are permitted.
4. Treatment with ultraviolet (UV) light (including tanning) during the 3 weeks prior to inclusion in this study.
5. Acute dermatitis outbreak or dermatitis on or near the test area on the back.
6. Conditions such as; fibromyalgia, chronic fatigue, depression, cognitive impairment, flu-like symptoms, diarrhea and/or headache without at least one of the symptoms related to metal exposure listed in Section 10.1 under physical examination
7. Inability to comply with patch test study requirements including multiple return visits and activity restrictions (e.g., protecting test panels from excess moisture due to showering or vigorous activity).
8. Participation in a clinical trial of an investigational drug, treatment or device during this study or 3 weeks prior to inclusion in this study.
9. An opinion of the Investigator that deems the potential subject to be non-compliant, unable to return for study visits or complete the study as detailed in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia L Norris, MD, Principal Investigator — Oregon Health & Science University, Portland USA; Karin Pacheco, MD, Principal Investigator — National Jewish Health School of Medicine, Colorado USA; Andreas Bircher, MD, Principal Investigator — University Hospital, Basel, Switzerland; Paolo Pigatto, MD, Principal Investigator — University of Milano, Italy; Thomas Rustemeyer, MD, PhD, Principal Investigator — VU University Medical Center, Netherlands; Peter Thomas, MD, Principal Investigator — Ludwig-Maximilians-Universität München, Germany; Maki Hosoki, DDS, PhD, Principal Investigator — Tokushima University Graduate School, Japan; Risa Tamagawa-Mineoka, MD, Principal Investigator — Kyoto Prefectural University of Medicine, Japan; Akiko Yagami, MD, PhD, Principal Investigator — Fujita Health University School of Medicine, Japan
Locations (8):
- National Jewish Health, University of Colorado Denver, Denver, Colorado, United States
- Ludwig-Maximilians-Universitat Munchen, Munich, Germany
- University of Milano, Milan, Italy
- Japan (3):
  - Fujita Health University School of Medicine, Aichi
  - Kyoto Prefectural University of Medicine, Kyoto
  - Tokushima University Graduate School, Tokushima
- VU University Medical Center, Amsterdam, Netherlands
- University Hospital Basel Allergology Unit, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study population will consist of subjects with past positive patch test result to at least one of the dilution series metals being tested on this study or strong suspicion of metal contact allergy.
Pre-assignment Details: Subjects with a past positive patch test will be tested with the allergen panel and corresponding reference allergen(s) to which they had the previous response. Subjects with suspicion of metal contact allergy will be tested with all dilution series and reference allergens. Not all subjects tested all allergens
Groups:
- All Subjects: All enrolled subjects were patch tested with ascending doses of investigational allergens on panes 1-5. At least 15 subjects with positive patch test responses (score of 1+, 2+ or 3+) were needed to determine optimal dose.
Period: Overall Study
Arm/Group | All Subjects
Started | 122
Completed | 121
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Baseline population: Enrolled subjects
Arm/Group | All Subjects
Number analyzed (Participants) | 122
Age, Continuous [Median (Full Range); unit: years] | 60.0 [26 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93
  Male | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 44
  European | 64
  Latin/South American/Caribbean | 1
  North American | 13
Region of Enrollment [Number; unit: participants]
  Netherlands | 20
  United States | 13
  Japan | 44
  Italy | 9
  Switzerland | 6
  Germany | 30
Subjects with past allergic response or suspicion of allergy [Count of Participants; unit: Participants] | 122

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Patch Test Responses
Description: Allergen patch test sites were scored at Visit 3 (day 3-4) Visit 4 (day 7-8) Visit 5 (day 10-14) and Visit 6 Day 19-23). Determination of positive or negative test response for each allergen dose was assessed by the investigator following the final visit.
Time Frame: 21 days post patch application
Population: Not all subjects tested all panels. No of subjects testing each panel; Panel 1- 105, Panel 2-111, Panel 3- 104, Panel 4- 109, Panel 5- 106
Measure: Count of Participants; unit: Participants
Groups:
- All Subjects: All enrolled subjects were patch tested with ascending doses of investigational allergens and excipient controls on panels 1-6. At least 15 subjects with positive patch test responses (score of 1+, 2+ or 3+) were needed to determine optimal dose. Allergen response pattern included number of positive responses that were late (initially observed at day 7 or later) or persistent (positive response that persisted from one study visit to the next) and number of negative responses that were doubtful or irritant.
Arm/Group | All Subjects
Number analyzed (Participants) | 121
Participants
  0.40 mg/cm2 aluminum chloride: Number Positive | 0
  0.40 mg/cm2 aluminum chloride: Number Negative | 105
  0.40 mg/cm2 aluminum chloride: Number not tested | 16
  0.12 mg/cm2 alumunum chloride: Number Positive | 0
  0.12 mg/cm2 alumunum chloride: Number Negative | 105
  0.12 mg/cm2 alumunum chloride: Number not tested | 16
  0.36 mg/cm2 aluminum chloride: Number Positive | 1
  0.36 mg/cm2 aluminum chloride: Number Negative | 104
  0.36 mg/cm2 aluminum chloride: Number not tested | 16
  0.72 mg/cm2 aluminum chloride: Number Positive | 4
  0.72 mg/cm2 aluminum chloride: Number Negative | 101
  0.72 mg/cm2 aluminum chloride: Number not tested | 16
  0.047 mg/cm2 aluminum lactate: Number Positive | 0
  0.047 mg/cm2 aluminum lactate: Number Negative | 105
  0.047 mg/cm2 aluminum lactate: Number not tested | 16
  0.14 mg/cm2 aluminum lactate: Number Positive | 0
  0.14 mg/cm2 aluminum lactate: Number Negative | 105
  0.14 mg/cm2 aluminum lactate: Number not tested | 16
  0.42 mg/cm2 aluminum lactate: Number Positive | 0
  0.42 mg/cm2 aluminum lactate: Number Negative | 105
  0.42 mg/cm2 aluminum lactate: Number not tested | 16
  0.84 mg/cm2 aluminum lactate: Number Positive | 0
  0.84 mg/cm2 aluminum lactate: Number Negative | 105
  0.84 mg/cm2 aluminum lactate: Number not tested | 16
  0.013 mg/cm2 copper sulfate: Number Positive | 2
  0.013 mg/cm2 copper sulfate: Number Negative | 109
  0.013 mg/cm2 copper sulfate: Number not tested | 10
  0.040 mg/cm2 copper sulfate: Number Positive | 9
  0.040 mg/cm2 copper sulfate: Number Negative | 102
  0.040 mg/cm2 copper sulfate: Number not tested | 10
  0.80 mg/cm2 copper sulfate: Number Positive | 10
  0.80 mg/cm2 copper sulfate: Number Negative | 101
  0.80 mg/cm2 copper sulfate: Number not tested | 10
  0.12 mg/cm2 copper sulfate: Number Positive | 16
  0.12 mg/cm2 copper sulfate: Number Negative | 95
  0.12 mg/cm2 copper sulfate: Number not tested | 10
  0.013 mg/cm2 manganese chloride: Number Positive | 1
  0.013 mg/cm2 manganese chloride: Number Negative | 103
  0.013 mg/cm2 manganese chloride: Number not tested | 17
  0.040 mg/cm2 manganese chloride: Number Positive | 0
  0.040 mg/cm2 manganese chloride: Number Negative | 103
  0.040 mg/cm2 manganese chloride: Number not tested | 18
  0.080 mg/cm2 manganese chloride: Number Positive | 4
  0.080 mg/cm2 manganese chloride: Number Negative | 99
  0.080 mg/cm2 manganese chloride: Number not tested | 18
  0.24 mg/cm2 manganese chloride: Number Positive | 29
  0.24 mg/cm2 manganese chloride: Number Negative | 74
  0.24 mg/cm2 manganese chloride: Number not tested | 18
  0.0067 mg/cm2 ammonium molybdate: Number Positive | 1
  0.0067 mg/cm2 ammonium molybdate: Number Negative | 103
  0.0067 mg/cm2 ammonium molybdate: Number not tested | 17
  0.02 mg/cm2 ammonium molybdate: Number Positive | 0
  0.02 mg/cm2 ammonium molybdate: Number Negative | 104
  0.02 mg/cm2 ammonium molybdate: Number not tested | 17
  0.040 mg/cm2 ammonium molybdate: Number Positive | 0
  0.040 mg/cm2 ammonium molybdate: Number Negative | 103
  0.040 mg/cm2 ammonium molybdate: Number not tested | 18
  0.12 mg/cm2 ammonium molybdate: Number Positive | 0
  0.12 mg/cm2 ammonium molybdate: Number Negative | 103
  0.12 mg/cm2 ammonium molybdate: Number not tested | 18
  0.0018 mg.cm2 tin chloride: Number Positive | 1
  0.0018 mg.cm2 tin chloride: Number Negative | 110
  0.0018 mg.cm2 tin chloride: Number not tested | 10
  0.037 mg/cm2 tin chloride: Number Positive | 4
  0.037 mg/cm2 tin chloride: Number Negative | 107
  0.037 mg/cm2 tin chloride: Number not tested | 10
  0.11 mg/cm2 tin chloride: Number Positive | 25
  0.11 mg/cm2 tin chloride: Number Negative | 86
  0.11 mg/cm2 tin chloride: Number not tested | 10
  0.33 mg/cm2 tin chloride: Number Positive | 65
  0.33 mg/cm2 tin chloride: Number Negative | 45
  0.33 mg/cm2 tin chloride: Number not tested | 11
  0.055 mg Ti/cm2 titanium citrate: Number Positive | 1
  0.055 mg Ti/cm2 titanium citrate: Number Negative | 108
  0.055 mg Ti/cm2 titanium citrate: Number not tested | 12
  0.11 mg Ti/cm2 titanium citrate: Number Positive | 2
  0.11 mg Ti/cm2 titanium citrate: Number Negative | 107
  0.11 mg Ti/cm2 titanium citrate: Number not tested | 12
  0.22 mg Ti/cm2 titanium citrate: Number Positive | 2
  0.22 mg Ti/cm2 titanium citrate: Number Negative | 106
  0.22 mg Ti/cm2 titanium citrate: Number not tested | 13
  0.07 mg Ti/cm2 titanium lactate: Number Positive | 2
  0.07 mg Ti/cm2 titanium lactate: Number Negative | 107
  0.07 mg Ti/cm2 titanium lactate: Number not tested | 12
  0.14 mg Ti/cm2 titanium lactate: Number Positive | 2
  0.14 mg Ti/cm2 titanium lactate: Number Negative | 107
  0.14 mg Ti/cm2 titanium lactate: Number not tested | 12
  0.28 mg Ti/cm2 titanium lactate: Number Positive | 4
  0.28 mg Ti/cm2 titanium lactate: Number Negative | 105
  0.28 mg Ti/cm2 titanium lactate: Number not tested | 12
  0.060 mg Ti/cm2 potassium titanium oxide oxalate: Number Positive | 1
  0.060 mg Ti/cm2 potassium titanium oxide oxalate: Number Negative | 108
  0.060 mg Ti/cm2 potassium titanium oxide oxalate: Number not tested | 12
  0.12 mg Ti/cm2 potassium titanium oxide oxalate: Number Positive | 5
  0.12 mg Ti/cm2 potassium titanium oxide oxalate: Number Negative | 104
  0.12 mg Ti/cm2 potassium titanium oxide oxalate: Number not tested | 12
  0.24 mg Ti/cm2 potassium titanium oxide oxalate: Number Positive | 2
  0.24 mg Ti/cm2 potassium titanium oxide oxalate: Number Negative | 107
  0.24 mg Ti/cm2 potassium titanium oxide oxalate: Number not tested | 12
  0.055 mg Ti/cm2 ammonium titanium oxide oxalate: Number Positive | 13
  0.055 mg Ti/cm2 ammonium titanium oxide oxalate: Number Negative | 96
  0.055 mg Ti/cm2 ammonium titanium oxide oxalate: Number not tested | 12
  0.11 mg Ti/cm2 ammonium titanium oxide oxalate: Number Positive | 21
  0.11 mg Ti/cm2 ammonium titanium oxide oxalate: Number Negative | 88
  0.11 mg Ti/cm2 ammonium titanium oxide oxalate: Number not tested | 12
  0.22 mg Ti/cm2 ammonium titanium oxide oxalate: Number Positive | 18
  0.22 mg Ti/cm2 ammonium titanium oxide oxalate: Number Negative | 91
  0.22 mg Ti/cm2 ammonium titanium oxide oxalate: Number not tested | 12
  0.0042 mg V/cm2 vanadium chloride: Number Positive | 0
  0.0042 mg V/cm2 vanadium chloride: Number Negative | 106
  0.0042 mg V/cm2 vanadium chloride: Number not tested | 15
  0.0083 mg V/cm2 vanadium chloride: Number Positive | 4
  0.0083 mg V/cm2 vanadium chloride: Number Negative | 102
  0.0083 mg V/cm2 vanadium chloride: Number not tested | 15
  0.025 mg V/cm2 vanadium chloride: Number Positive | 25
  0.025 mg V/cm2 vanadium chloride: Number Negative | 81
  0.025 mg V/cm2 vanadium chloride: Number not tested | 15
  0.050 mg V/cm2 vanadium chloride: Number Positive | 46
  0.050 mg V/cm2 vanadium chloride: Number Negative | 60
  0.050 mg V/cm2 vanadium chloride: Number not tested | 15
  0.0042 mg V/cm2 vanadium sulfate: Number Positive | 6
  0.0042 mg V/cm2 vanadium sulfate: Number Negative | 100
  0.0042 mg V/cm2 vanadium sulfate: Number not tested | 15
  0.0083 mg V/cm2 vanadium sulfate: Number Positive | 7
  0.0083 mg V/cm2 vanadium sulfate: Number Negative | 99
  0.0083 mg V/cm2 vanadium sulfate: Number not tested | 15
  0.025 mg V/cm2 vanadium sulfate: Number Positive | 10
  0.025 mg V/cm2 vanadium sulfate: Number Negative | 96
  0.025 mg V/cm2 vanadium sulfate: Number not tested | 15
  0.050 mg V/cm2 vanadium sulfate: Number Positive | 30
  0.050 mg V/cm2 vanadium sulfate: Number Negative | 76
  0.050 mg V/cm2 vanadium sulfate: Number not tested | 15
  0.013 mg/cm2 zinc chloride: Number Positive | 2
  0.013 mg/cm2 zinc chloride: Number Negative | 109
  0.013 mg/cm2 zinc chloride: Number not tested | 10
  0.040 mg/cm2 zinc chloride: Number Positive | 7
  0.040 mg/cm2 zinc chloride: Number Negative | 104
  0.040 mg/cm2 zinc chloride: Number not tested | 10
  0.080 mg/cm2 zinc chloride: Number Positive | 13
  0.080 mg/cm2 zinc chloride: Number Negative | 98
  0.080 mg/cm2 zinc chloride: Number not tested | 10
  0.24 mg/cm2 zinc chloride: Number Positive | 69
  0.24 mg/cm2 zinc chloride: Number Negative | 42
  0.24 mg/cm2 zinc chloride: Number not tested | 10
Statistical Analysis 1: Comparison: All Subjects; Comparison between 0.12 mg/cm2 copper sulfate and copper sulfate 2% in petrolatum; Test type: Other; Kappa statistic = 0.28, 95% CI 2-sided [-0.01 to 0.58]
Statistical Analysis 2: Comparison: All Subjects; Comparison between 0.24 mg/cm2 manganese chloride and manganese chloride 2% in petrolatum; Test type: Other; Kappa statistic = 0.45, 95% CI 2-sided [0.24 to 0.66]
Statistical Analysis 3: Comparison: All Subjects; Comparison between 0.33 mg/cm2 tin chloride and tin chloride 1% in petrolatum; Test type: Other; Kappa statistic = 0.23, 95% CI 2-sided [0.07 to 0.38] — Kappa statistic is for 0.33 mg/cm2 tin chloride vs 1% tin chloride in petrolatum reference allergen
Statistical Analysis 4: Comparison: All Subjects; Comparison between 0.22 mg Ti/cm2 ammonium titanium oxide oxalate and ammnium titanium oxide oxalate 19% in petrolatum; Test type: Other; Kappa statistic = 0.40, 95% CI 2-sided [0.15 to 0.65] — Kappa statistic is for 0.22 mg Ti/cm2 ammonium titanium oxide oxalate vs 19% ammonium titanium oxide oxalate in petrolatum reference allergen
Statistical Analysis 5: Comparison: All Subjects; Comparison between 0.050 mg/cm2 vanadium sulfate and vanadium sulfate 1.5% in petrolatum; Test type: Other; Kappa statistic = 0.52, 95% CI 2-sided [0.30 to 0.73] — Kappa statistic is for 0.050 mg V/cm2 vanadium sulfate vs 1.5% vanadium sulfate in petrolatum reference allergen
Statistical Analysis 6: Comparison: All Subjects; Comparison betweenm 0.24 mg/cm2 zinc chloride and zinc chloride 2% in petrolatum; Test type: Other; Kappa statistic = 0.36, 95% CI 2-sided [0.07 to 0.38] — Kappa statistic is for 0.24 mg/cm2 zinc chloride vs 2% zinc chloride in petrolatum reference allergen

2. Secondary Outcome: Number of Subjects With Panel Adhesion
Description: Panel Adhesion was measured at Visit 2 (day 2) prior to panel removal according to the following scale: Excellent- Skin contact good; all tape edges adherent; all allergens in contact with the skin, Good- Skin contact acceptable; some tape edges lifting; all allergens in contact with the skin, Poor- Little to no skin contact with panel; one or more allergens not in contact with the skin, Detached- Panel completely off the skin; none of the allergens in contact with the skin
Time Frame: Day 2, visit 2 prior to panel removal
Measure: Count of Participants; unit: Participants
Groups:
- All Subjects: All enrolled subjects were patch tested with ascending doses of investigational allergens and excipient controls on panels 1-6. At least 15 subjects with positive patch test responses (score of 1+, 2+ or 3+) were needed to determine optimal dose.
Arm/Group | All Subjects
Number analyzed (Participants) | 121
Participants
  Panel 1 Adhesion: Excellent | 102
  Panel 1 Adhesion: Good | 1
  Panel 1 Adhesion: Poor | 2
  Panel 1 Adhesion: Detached | 0
  Panel 1 Adhesion: Not Tested | 16
  Panel 2 Adhesion: Excellent | 103
  Panel 2 Adhesion: Good | 3
  Panel 2 Adhesion: Poor | 5
  Panel 2 Adhesion: Detached | 0
  Panel 2 Adhesion: Not Tested | 10
  Panel 3 Adhesion: Excellent | 98
  Panel 3 Adhesion: Good | 3
  Panel 3 Adhesion: Poor | 3
  Panel 3 Adhesion: Detached | 0
  Panel 3 Adhesion: Not Tested | 17
  Panel 4 Adhesion: Excellent | 105
  Panel 4 Adhesion: Good | 1
  Panel 4 Adhesion: Poor | 3
  Panel 4 Adhesion: Detached | 0
  Panel 4 Adhesion: Not Tested | 12
  Panel 5 Adhesion: Excellent | 100
  Panel 5 Adhesion: Good | 6
  Panel 5 Adhesion: Poor | 0
  Panel 5 Adhesion: Detached | 0
  Panel 5 Adhesion: Not Tested | 15
  Panel 6 Adhesion: Excellent | 113
  Panel 6 Adhesion: Good | 5
  Panel 6 Adhesion: Poor | 2
  Panel 6 Adhesion: Detached | 0
  Panel 6 Adhesion: Not Tested | 1

3. Secondary Outcome: Tape Irritation
Description: Tape irritation was measured according to the following scale: None- No irritation, Weak- Faint to definite pink erythema, Moderate- Moderate erythema, definite redness, Strong- Severe erythema, very intense redness. Following visit 6, the Investigators rated tape irritation based on the overall trend observed at visits 2-6. Irritation at visit 2 that resolved by visit 3 was considered none. Skin under occlusion from an adhesive material would be expected to have minimal irritation shortly after the panel is removed. Irritation that persisted or increased in severity beyond visit 3 but resolved by the following visit would have been rated as irritant. An allergic response was considered if irritation persisted beyond visit 3, increased in severity and had symptoms consistent with criteria used to score positive skin reactions according to standard patch testing guidelines established by the International Contact Dermatitis Research Group.
Time Frame: Visit 2 (day 2), visit 3 (day 3-4), visit 4 (day 7-8) visit 5 (day 10-14), visit 6 (day 19-23) with overall assessment by the Investigator following visit 6
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 121
Participants
  Panel 1 Tape Irritation: None | 103
  Panel 1 Tape Irritation: Irritant | 2
  Panel 1 Tape Irritation: Allergic | 0
  Panel 1 Tape Irritation: Not Tested | 16
  Panel 2 Tape Irritation: None | 109
  Panel 2 Tape Irritation: Irritant | 2
  Panel 2 Tape Irritation: Allergic | 0
  Panel 2 Tape Irritation: Not Tested | 10
  Panel 3 Tape Irritation: None | 103
  Panel 3 Tape Irritation: Irritant | 1
  Panel 3 Tape Irritation: Allergic | 0
  Panel 3 Tape Irritation: Not Tested | 17
  Panel 4 Tape Irritation: None | 108
  Panel 4 Tape Irritation: Irritant | 1
  Panel 4 Tape Irritation: Allergic | 0
  Panel 4 Tape Irritation: Not Tested | 12
  Panel 5 Tape Irritation: None | 105
  Panel 5 Tape Irritation: Irritant | 1
  Panel 5 Tape Irritation: Allergic | 0
  Panel 5 Tape Irritation: Not Tested | 15
  Panel 6 Tape Irritation: None | 119
  Panel 6 Tape Irritation: Irritant | 1
  Panel 6 Tape Irritation: Allergic | 0
  Panel 6 Tape Irritation: Not Tested | 1

4. Secondary Outcome: Chip Irritation
Description: Chip irritation was measured according to the following scale: None- No irritation, Weak- Faint to definite pink erythema, Moderate- Moderate erythema, definite redness, Strong- Severe erythema, very intense redness. Following visit 6, the Investigators rated Chip irritation based on the overall trend observed at visits 2-6. Irritation at visit 2 that resolved by visit 3 was considered none. Skin under occlusion from an adhesive material would be expected to have minimal irritation shortly after the panel is removed. Irritation that persisted or increased in severity beyond visit 3 but resolved by the following visit would have been rated as irritant. An allergic response was considered if irritation persisted beyond visit 3, increased in severity and had symptoms consistent with criteria used to score positive skin reactions according to standard patch testing guidelines established by the International Contact Dermatitis Research Group.
Time Frame: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 121
Participants
  Panel 1 Chip Irritation: None | 105
  Panel 1 Chip Irritation: Irritant | 0
  Panel 1 Chip Irritation: Allergic | 0
  Panel 1 Chip Irritation: Not Tested | 16
  Panel 2 Chip Irritation: None | 111
  Panel 2 Chip Irritation: Irritant | 0
  Panel 2 Chip Irritation: Allergic | 0
  Panel 2 Chip Irritation: Not Tested | 10
  Panel 3 Chip Irritation: None | 104
  Panel 3 Chip Irritation: Irritant | 0
  Panel 3 Chip Irritation: Allergic | 0
  Panel 3 Chip Irritation: Not Tested | 17
  Panel 4 Chip Irritation: None | 109
  Panel 4 Chip Irritation: Irritant | 0
  Panel 4 Chip Irritation: Allergic | 0
  Panel 4 Chip Irritation: Not Tested | 12
  Panel 5 Chip Irritation: None | 106
  Panel 5 Chip Irritation: Irritant | 0
  Panel 5 Chip Irritation: Allergic | 0
  Panel 5 Chip Irritation: Not Tested | 15
  Panel 6 Chip Irritation: None | 120
  Panel 6 Chip Irritation: Irritant | 0
  Panel 6 Chip Irritation: Allergic | 0
  Panel 6 Chip Irritation: Not Tested | 1

ADVERSE EVENTS:
Time Frame: Day 2-21
Description: Because subjects were patched with multiple allergens/doses it is not possible to relate adverse events to a single allergen/dose
Groups:
- All Subjects: Subjects patched with at least 1 patch test panel were included in adverse event reporting.
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 0/122
Serious Adverse Events (participants affected / at risk) | 1/122
Other Adverse Events (participants affected / at risk) | 30/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=122)
Ductal carcinoma of right breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=122)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Hordeolum (Eye disorders) | 1 (1)
Abdominal pain, upper (Gastrointestinal disorders) | 1 (1)
Glossitis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Periodontal inflammation (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Application site erythema (General disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Inflammation (General disorders) | 1 (1)
Influenza-like illness (General disorders) | 2 (2)
Malaise (General disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Cystitis (Infections and infestations) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 3 (3)
Tension headache (Nervous system disorders) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Endodontic tooth pain (Surgical and medical procedures) | 1 (1)
Therapeutic nerve ablation (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-06-27): https://cdn.clinicaltrials.gov/large-docs/49/NCT02615249/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-30): https://cdn.clinicaltrials.gov/large-docs/49/NCT02615249/SAP_001.pdf